CLINICAL TRIAL: NCT04022694
Title: Preventing Non-communicable Diseases in Guatemala Through Sugary Drink Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Universidad Rafael Landivar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21TW010837 (NIH); R21TW010837 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Food Preferences
Keywords: Food Labeling; Adolescents
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Three private schools will be enrolled in the study (two larger, one smaller) that have students between the ages of 12 and 18. There will be no posters displayed at any of the schools during the baseline period. The two larger schools will be randomized to either an SSB warning/non-SSB promoting poster or a calorie/control poster that will be implemented in the school cafeterias during a four-week intervention period. To increase the sample size for the intervention condition, the intervention will also be implemented at a smaller school. For the primary analysis, data only from schools that were randomized to condition will be used. Data was collected from both a sample of participants & from the cash registers directly.
Masking Description: Participants will be told the researchers are interested in cafeteria purchase preferences, but participants will not know which condition has been assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie/Control Poster (Active Comparator): This poster will display images of both SSBs and low or no sugar beverages with calories listed below the beverages. It will simply state that those beverages are sold in the school store.
  Interventions: Behavioral: Exposure to beverage calorie information
- SSB Warning and Non-SSB Promotion Poster (Experimental): This poster will display images of both SSBs and low or no sugar beverages with calories listed below the beverages. In addition, the message will state that SSBs are high in sugar and should be avoided, while low or no sugar beverages are healthier options and should be chosen.
  Interventions: Behavioral: Exposure to beverage health information; Behavioral: Exposure to beverage calorie information
- Baseline for Calorie/Control Poster (No Intervention): We will collect baseline data from a group of students before posting the Calorie/Control Poster in the control school.
- Baseline for SSB Warning and Non-SSB Promotion Poster (No Intervention): We will collect baseline data from a group of students before posting the SSB Warning and Non-SSB Promotion Poster in the intervention school.

INTERVENTIONS:
Behavioral: Exposure to beverage health information — Red stop sign and avoidance message for sugar-sweetened beverages and green check mark and promotion message for non-sugar-sweetened beverage nutrition information
  Arms: SSB Warning and Non-SSB Promotion Poster
Behavioral: Exposure to beverage calorie information — Calories for sugar-sweetened and non-sugar-sweetened beverages
  Arms: Calorie/Control Poster; SSB Warning and Non-SSB Promotion Poster

SUMMARY:
Sugar-sweetened beverages are a significant contributor to adult and childhood obesity in Guatemala. Policies to place health warning labels on sugar-sweetened beverages are being pursued, but there is little empirical data on how such labels influence people. The primary aim of this study is to test the association between sugar-sweetened beverage (SSB) warning posters compared to control posters and change in SSBs purchased compared to baseline by adolescents shopping at school cafeterias in Guatemala City, Guatemala. The hypothesis is that posters with information warning people of the health harms associated with overconsuming SSBs and promoting low sugar beverages will be associated with greater reductions in SSB purchases compared to a control poster.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 18 years old
* Made a food or beverage purchase
* Has permission from parent or caregiver to participate
* Has not yet completed the purchase assessment

Exclusion Criteria:

* Under 12 or over 18 years old
* Did not make a food or beverage purchase
* Parent or caregiver refused to give child permission to participate
* Already participated in the purchase assessment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 628 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Universidad Rafael Landivar, Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We do not report data from 166 participants collected at a 3rd smaller school because that school was assigned (not randomized) to the SSB Warning and Non-SSB Promotion Poster because of its smaller size.
Groups:
- Calorie/Control Poster: This poster will display images of both Sugar Sweetened Beverages (SSBs) and low or no sugar beverages with calories listed below the beverages. It will simply state that those beverages are sold in the school store.
  Exposure to beverage calorie information: Calories for sugar-sweetened and non-sugar-sweetened beverages
- SSB Warning and Non-SSB Promotion Poster: This poster will display images of both Sugar Sweetened Beverages (SSBs) and low or no sugar beverages with calories listed below the beverages. In addition, the message will state that SSBs are high in sugar and should be avoided, while low or no sugar beverages are healthier options and should be chosen.
  Exposure to beverage health information: Red stop sign and avoidance message for sugar-sweetened beverages and green check mark and promotion message for non-sugar-sweetened beverage nutrition information
  Exposure to beverage calorie information: Calories for sugar-sweetened and non-sugar-sweetened beverages
Period: Overall Study
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Started | 167 | 145 | 143 (This was a cross-sectional study, so participants at baseline -- were not the same as exposure.) | 173 (This was a cross-sectional study, so participants at baseline -- were not the same as exposure.)
Completed | 167 | 145 | 143 | 173
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data on race was not collected for participants assigned to the Arms/Groups "Calorie/Control Poster" and "SSB Warning and Non-SSB Promotion Poster" because these data were collected in Guatemala and race would have a different meaning than race in the United States.
Groups:
- Baseline for SSB Warning and Non-SSB Promotion Poster: We will collect baseline data from a group of students before posting the SSB Warning and Non-SSB Promotion Poster in the treatment school.
- Total: Total of all reporting groups
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Total
Number analyzed (Participants) | 167 | 145 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 167 | 145 | 312
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.6) | 14.9 (1.4) | 15.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 68 | 126
  Male | 109 | 77 | 186
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Guatemala | 167 | 145 | 312

OUTCOME MEASURES:

1. Primary Outcome: Volume of SSBs Per Transaction
Description: Total milliliters of SSBs per transaction from sales data
Time Frame: Through study period (either 4 weeks baseline, or 4 weeks intervention)
Population: In addition to the surveys with the participants (described in the participant flow), data on total sales were collected at the register. It is not possible to know if these sales data were associated with one or more than one participant because they are at the sales item level. For the purposes of this report, the number of participants are identical to the number of items sold.
Measure: Mean (Standard Deviation); unit: mL of Sugar Sweetened Beverages purchase
Units Other Than Participants: sales item
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (sales item) | 3642 | 3477 | 3898 | 3533
mL of Sugar Sweetened Beverages purchase | 116.2 (212.5) | 89.8 (160.1) | 115.3 (211.8) | 103.4 (176.2)

2. Primary Outcome: Beverage Calories Per Transaction
Description: Total number of calories for all beverages (SSBs and non-SSBs) per transaction from sales data
Time Frame: Through study period (either 4 weeks baseline or 4 weeks intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beverage calories sold
Units Other Than Participants: sales item
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (sales item) | 3642 | 3477 | 3898 | 3533
beverage calories sold | 45.1 (83.7) | 35.9 (67.1) | 41.2 (75.9) | 39.0 (69.0)

3. Secondary Outcome: Total Calories Per Transaction
Description: Total number of calories for all food and beverages (SSBs and non-SSBs) per transaction from purchase assessments (e.g., calories from Coke + bag of chips)
Time Frame: Through time frame (either 4 weeks baseline, or 4 weeks intervention)
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 167 | 145 | 143 | 173
calories | 290.8 (224.2) | 338.5 (222.6) | 287.5 (211.8) | 332.0 (239.8)

4. Other Pre Specified Outcome: Percentage of Participants With Transactions With SSBs Out of All Food and Beverage Transactions
Description: Percentage of participants with transactions that have sugar sweetened beverages out of all participants who had food and beverage transactions
Time Frame: 4-week baseline and 4-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 167 | 145 | 143 | 173
Participants | 57 | 36 | 40 | 63

5. Other Pre Specified Outcome: Percentage of Participants With Transactions With SSBs Out of All Beverage Transactions
Description: Percentage of participants with transactions that have sugar sweetened beverages out of all participants who had beverage transactions
Time Frame: 4-week baseline and 4-week intervention
Population: This analysis was limited to people who bought a beverage. Students who only purchased food were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 76 | 65 | 48 | 105
Participants | 57 | 36 | 40 | 63

6. Other Pre Specified Outcome: Unhealthy Perceptions of SSBs
Description: Average of perceptions of healthiness (measured on Likert scales) for two items (1=Extremely unhealthy; 7=Extremely healthy, lower values are more accurate)
Time Frame: 4 weeks baseline, 4 weeks intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 167 | 145 | 143 | 173
units on a scale | 3.05 (1.07) | 3.04 (0.98) | 3.09 (1.06) | 3.02 (1.00)

7. Other Pre Specified Outcome: Healthy Perceptions of Non-SSBs
Description: Average of perceptions of healthiness (measured on Likert scales) for two items (1=Extremely unhealthy; 7=Extremely healthy, higher values are more accurate)
Time Frame: 4 weeks baseline, 4 weeks intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 167 | 145 | 143 | 173
units on a scale | 4.79 (0.81) | 4.83 (0.77) | 5.01 (0.87) | 4.96 (0.79)

8. Other Pre Specified Outcome: Perceived Influence of Poster Among Those Who Saw it
Description: "Do you think the poster influenced what you purchased?" (1=Not at all; 5=Very much, higher values in the intervention condition indicate the intervention is perceived to be effective)
Time Frame: During intervention, 4 weeks
Population: Only asked in the treatment period of participants who reported seeing a poster.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 87 | 110
units on a scale | 2.01 (1.25) | 2.51 (1.36)

9. Other Pre Specified Outcome: Poster Message Trust
Description: "How much do you trust the information on the poster?" (1=Not at all; 5=Very much, higher values in the intervention condition indicate the intervention is perceived to be trustworthy)
Time Frame: During intervention, 4 weeks
Population: Only asked during the intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
Number analyzed (Participants) | 143 | 173
units on a scale | 3.55 (1.16) | 3.94 (0.86)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Baseline for Calorie/Control Poster | Baseline for SSB Warning and Non-SSB Promotion Poster | Calorie/Control Poster | SSB Warning and Non-SSB Promotion Poster
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/145 | 0/143 | 0/173
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/145 | 0/143 | 0/173
Other Adverse Events (participants affected / at risk) | 0/167 | 0/145 | 0/143 | 0/173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT04022694/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT04022694/SAP_001.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT04022694/ICF_002.pdf